CLINICAL TRIAL: NCT07359001
Title: Development of Video-based Sit-to-stand Evaluation Tool for Stroke Patients
Brief Title: Video-based Sit-to-stand Evaluation for Stroke Patients
Status: Completed | Type: Observational
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hanbin Kim, PhD Student, Sahmyook University
Other Study IDs: SYU 2022-10-012-007
Record Dates: First submitted 2025-11-27; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Stroke Rehabilitation
Keywords: Stroke; Telerehabilitation; Scale; Reproducibility of Results; Correlation of Data; Biomechanical Phenomena; Range of Motion, Articular; Video Recording; Posture
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: No interventions are provided. They will be video recorded during their sit-to-stand trials of three
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Stroke patients are video recorded during three sit-to-stand trials with 5 minutes rest between the trials.

SUMMARY:
The purpose of this study is to develop and validate a novel video-based postural evaluation tool designed to objectively measure the quality and dynamics of the Sit-to-Stand (STS) motion in stroke patients, specifically allowing physical therapists to monitor patient progress remotely via tele-evaluation. Since stroke survivors often face difficulties attending regular in-clinic assessments, this tool addresses a critical unmet need. The core question this study aims to answer is whether this new video-based measurement can accurately and consistently assess standing ability when compared against established standards. To confirm the tool's trustworthiness, we will first test its reliability by assessing if different experts achieve the same results (Inter-rater reliability) and if the same expert achieves the same results across multiple trials (Intra-rater reliability). We will then confirm the tool's accuracy (validity) by examining if its derived scores correlate strongly with established clinical measures (e.g., Trunk Impairment Scale, TIS) and patient-reported outcome measures. Finally, we will verify its scientific precision by comparing the tool's detailed kinematic measurements (including total STS time and joint angles) against the gold-standard data derived from the Kinovea motion analysis software.

DETAILED DESCRIPTION:
1. Rationale and Context

   - Stroke remains a leading global cause of long-term functional disability. While early functional recovery is rapid, many patients require sustained long-term rehabilitation. Access to adequate rehabilitation is often compromised by geographical and institutional barriers, highlighting a critical unmet need in clinical practice. Tele-rehabilitation, utilizing Information and Communications Technology (ICT) via devices such as smartphones and tablets, is presented as a vital alternative to enhance accessibility and provide continuous, systematic care without the need for physical travel. The success of tele-rehabilitation fundamentally depends on the availability of assessment tools that can objectively and reliably measure functional changes from a distance.
2. Scientific Focus: Sit-to-Stand (STS) Movement

   - The Sit-to-Stand (STS) task is a foundational activity of daily living, demanding complex coordination of lower extremity strength, balance, posture control, and weight shifting. Post-stroke, patients exhibit significant limitations in STS due to asymmetric weight-bearing, decreased strength, and impaired postural control, which increases the risk of falls. Therefore, the assessment of STS must extend beyond simple quantitative measures (e.g., time or repetition counts, such as FTSTS or TUG) to capture the qualitative characteristics (e.g., symmetry, compensatory strategies) essential for guiding therapeutic intervention. This study addresses the current limitation of existing qualitative tools that require direct, in-person observation by developing a tool suitable for non-face-to-face video analysis.
3. Assessment Tool Development Methodology

   * The study utilized a multi-stage process for tool construction, ensuring both clinical relevance and theoretical soundness:
   * Initial Item Generation: The preliminary tool items were compiled based on a comprehensive literature review and clinical books related to stroke patient posture and balance assessment, with a specific focus on alignment and movement analysis during STS. The tool ultimately adopted concepts from Raine et al.'s Bobath concept theory.
   * Item Structuring: The STS movement was segmented into five functional phases (including a preparation phase added later). The items, totaling 29 items, are structured for observation from both the frontal and sagittal (affected side) planes, and scored on a 5-point Likert scale for most items.
   * Validation Procedures (Content/Face Validity): The preliminary tool underwent rigorous validation. Face validity was assessed by a panel of expert physical therapists. Content validity was verified by 10 neurological rehabilitation therapists with over 10 years of experience, following established procedures. This iterative process led to the deletion, modification, and addition of items, ensuring the tool's clinical relevance and comprehensiveness.
   * Video Recording Protocols: To minimize observational bias and establish remote feasibility, the assessment guidelines mandate that the STS movement be recorded from the patient's front (coronal view) and affected side (sagittal view). The videos are then edited to allow simultaneous viewing of both perspectives, ensuring full visibility from head to toe.
4. Study Procedures for Reliability

   * The final version of the tool was tested using video recordings of STS movements from 10 chronic stroke patients. The assessments were conducted by 10 neurological physical therapists with over three years of experience.
   * Inter-Rater Reliability: Measured the consistency of scoring among the 28 different evaluators using the same video recordings. The ICC(2,1) model was applied for this analysis.
   * Intra-Rater Reliability: Measured the consistency of individual evaluators by having the same 10 evaluators assess the identical video recordings two times, separated by an interval of approximately 6 months. The ICC(3,1) model was applied for this analysis.
5. Statistical Analysis The consistency of measurements (Reliability) was quantified using the Intraclass Correlation Coefficient (ICC). The interpretation of the ICC values followed standard guidelines (e.g., ICC ≥0.90 is considered 'excellent', 0.75-0.90 is 'good', 0.50-0.75 is 'moderate').

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stroke resulting in motor impairment.
* Patients in the chronic phase, defined as being more than one year post-diagnosis.
* Patients capable of performing the Sit-to-Stand (STS) movement independently without the use of walking aids or physical assistance.
* Patients who fully understand the study purpose and procedures and have voluntarily provided written informed consent.

Exclusion Criteria:

* Exclusion criteria included individuals with visual, auditory, or vestibular impairments, cognitive dysfunction, more than two episodes of stroke, or other neurological impairments.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of stroke patients currently admitted to H Hospital located in Namyangju-si, Gyeonggi-do, South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Inter-rater Reliability of the Video-Based Sit-to-Stand (STS) Assessment Tool as Assessed by the Intraclass Correlation Coefficient (ICC 2,1) | At baseline, during a single assessment session following enrollment
  The inter-rater reliability assesses the degree of agreement among 28 different physical therapists evaluating the same patient videos. The video-based STS assessment tool consists of 29 items across 5 phases (Phase 0: Preparation, Phase 1: Flexion Momentum, Phase 2: Momentum Transfer, Phase 3: Extension, Phase 4: Stabilization). Each item is scored on a 5-point Likert scale ranging from 1 (poor performance/unable) to 5 (perfect performance). The total score is the sum of all items. Reliability is reported using the Intraclass Correlation Coefficient (ICC) model 2,1. An ICC value ≥ 0.90 indicates excellent reliability, 0.75-0.90 good, 0.50-0.75 moderate, and < 0.50 poor reliability.
Intra-rater Reliability of the Video-Based Sit-to-Stand (STS) Assessment Tool as Assessed by the Intraclass Correlation Coefficient (ICC 3,1) | At baseline, during a single assessment session following enrollment
  The intra-rater reliability assesses the consistency of the same rater's scoring over time. Ten physical therapists evaluated the same patient video recordings at baseline and again after a specific interval. The assessment tool comprises 29 items scored on a 1 to 5 scale, where higher scores indicate better performance. The consistency between the two time points is calculated using the Intraclass Correlation Coefficient (ICC) model 3,1.

SECONDARY OUTCOMES:
Criterion Validity: Correlation Between the Video-Based STS Assessment Tool Score and the Trunk Impairment Scale (TIS) Score | At baseline, during a single assessment session following enrollment
  To establish criterion validity, the total score obtained from the newly developed video-based STS assessment tool is correlated with the score from the Trunk Impairment Scale (TIS). The TIS is a validated tool measuring static and dynamic sitting balance and trunk coordination. TIS scores range from 0 to 23, with higher scores indicating better trunk performance. A Pearson or Spearman correlation coefficient will be calculated to determine the strength of the relationship.
Criterion Validity: Correlation Between the Video-Based STS Assessment Tool Score and Total Sit-to-Stand Duration | At baseline, during a single assessment session following enrollment
  This measure establishes construct validity by analyzing the relationship between the qualitative assessment (video tool score) and the quantitative performance (speed). A correlation coefficient will be calculated between the total score obtained from the video-based assessment tool (range: 29-145, higher scores indicate better movement quality) and the total time (in seconds) required for the patient to complete the Sit-to-Stand task. This tests the hypothesis that better movement quality correlates with more efficient (faster) performance.
Construct Validity: Correlation Between Video-Based STS Assessment Tool Scores and Kinematic Parameters (Joint Angles and Angular Velocities) Measured by Kinovea Software | At baseline, during a single assessment session following enrollment
  To verify construct validity, the scores from the video-based tool are compared against quantitative motion analysis data obtained using Kinovea software. The specific kinematic parameters analyzed include the range of motion (degrees) and angular velocity (degrees/second) of the hip, knee, and ankle joints during the Sit-to-Stand motion. Correlation coefficients will be calculated to determine how well the video-based tool's qualitative scores reflect the objective kinematic changes measured by the software.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Science Hall 3, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided